CLINICAL TRIAL: NCT04637425
Title: The Effect of Polyvalent Mechanical Bacterial Lysate on the Reduction of Nasal Staphylococcus Aureus Carriage in Children With Pollen Allergic Rhinitis
Brief Title: Effect of Bacterial Lysate on Nasal Carriage of Staphylococcus Aureus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of Lublin (Other)
Responsible Party: Principal Investigator, Kamil Janeczek, Principal Investigator, Medical University of Lublin
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KE-0254/41/2018(2)
Record Dates: First submitted 2020-11-15; First posted 2020-11-19 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2020-12

CONDITIONS: Allergic Rhinitis
Keywords: allergic rhinitis; seasonal allergic rhinitis; children; grass pollen season; bacterial lysate; nasal Staphylococcus aureus carriage
MeSH Terms: conditions — Rhinitis, Allergic; Rhinitis, Allergic, Seasonal | interventions — Broncho-Vaxom

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ismigen (Experimental): Treatment over 3 successive months with one daily tablet over 10 days followed by 20 days of rest.
  Interventions: Drug: Ismigen
- Placebo (Placebo Comparator): Treatment over 3 successive months with one daily tablet over 10 days followed by 20 days of rest.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ismigen — Sublingual tablets containing 7 mg of bacterial lysate from the following bacteria: Staphylococcus aureus, Haemophilus influenzae serotype B, Klebsiella pneumoniae, Klebsiella ozaenae, Neiserria catarrhalis, Streptococcus viridans, Streptococcus pyogenes, Streptococcus pneumoniae (6 strains: TY1/EQ11, TY2/EQ22, TY3/EQ14, TY5/EQ15, TY8/EQ23, TY47/EQ24) - sublingual use 1 tablet per day over 10 days for 3 successive months.
  Other Names: Polyvalent Mechanical Bacterial Lysate (PMBL)
  Arms: Ismigen
Drug: Placebo — Matched tablets without any active substance.
  Arms: Placebo

SUMMARY:
This study assesses the effectiveness of Polyvalent Mechanical Bacterial Lysate (PMBL-Ismigen) in reducing nasal methicillin-resistant Staphylococcus aureus (MRSA) colony growth in children with pollen allergic rhinitis (AR) aged 5 to 17. Half of the participants received PMBL and the other half received a placebo.

DETAILED DESCRIPTION:
Seasonal allergic rhinitis (SAR) is caused by the allergens of wind-pollinated plants, and in Poland mainly by grass pollen allergens. During the grass pollen season, patients may suffer from fatigue, weakness, lack of fitness, difficulty in sleeping and reduced performance at school. In people allergic to the above-mentioned pollen, the disease significantly reduces the quality of life and requires intensive treatment in the pollen period.

MRSA colonizing the nasal cavity has the ability to actively modulate the immune response in children suffering from SAR. Many studies have shown a greater severity of AR symptoms in patients with a MRSA-positive nasal swab compared to patients with normal nasal flora.

Due to the high incidence of AR, the negative impact of the disease on the quality of life, and incomplete effectiveness of previously available therapeutic methods, new methods of treatment are being developed. Recent research highlights the immunoregulatory potential of bacterial lysates, indicating the possibility of their future use in the prevention and treatment of allergic diseases, including atopic dermatitis, AR, and asthma.

Based on the above considerations, it can be hypothesized that bacterial lysates reduce the severity of AR symptoms by eradicating MRSA from the nasal cavity. However, so far no randomized, double-blind, placebo-controlled study has been conducted to evaluate the effect of bacterial lysates on nasal Staphylococcus aureus carriage in children with SAR.

The main aim of this study was to evaluate nasal colonization by MRSA among children with SAR and the effect of PMBL on the reduction of MRSA colony growth in these children.

70 children with SAR were enrolled to this study and were randomly assigned to the PMBL group (n=35) and placebo group (n=35). Two visits took place as part of the study: at the beginning of the grass pollen season and at the end of the season. The time frame of the grass pollen season for south-eastern Poland was determined using the "95%" method on the basis of measurements of grass pollen concentration in the atmospheric air, which were obtained from the Environmental Allergy Research Centre in Warsaw. Nasal swabs for bacteriological cultures were taken at each visit and were transferred to the hospital laboratory.

ELIGIBILITY:
Inclusion Criteria:

* Children of both genders aged 5 to 17 years.
* Children with grass pollen-induced allergic rhinitis recognized and treated according to current ARIA (Allergic Rhinitis and its Impact on Asthma) recommendations.
* Positive skin prick test to grass pollen allergens or positive specific IgE (defined as ≥ class 2, ≥ 0,70 kU/l) against timothy grass pollen allergens.
* Presentation of clinical symptoms of the allergic rhinitis (rhinorrhea, nasal congestion, nasal itching, sneezing) in at least two recent grass pollen seasons in Poland before inclusion in the study.
* Proper use of polyvalent mechanical bacterial lysate sublingual tablets.
* Written informed consent obtained from parents/guardians before any study related procedures are performed.

Exclusion Criteria:

* Patient received mechanical or any other polyvalent bacterial lysate immunostimulation within the previous 12 months before randomisation visit.
* Patient received oral/subcutaneous allergen-immunotherapy within the previous 3 years before the start of the study.
* Vaccination performed within 3 months before the beginning of the study.
* Deficiencies in cellular and humoral immunity.
* Treatment with antibiotics within the last 1 month before the start of the study.
* Treatment with systemic corticosteroids within the last 6 months before the start of the study.
* Pregnant or breastfeeding woman.
* Other chronic conditions of the nose or nasal sinuses.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2018-04-22 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Change in the growth intensity of the nasal Staphylococcus aureus colony | at baseline, and at 3-months
  At the randomization visit and end-of-study visit, a nasal swab was collected for bacteriological cultures and compared whether there was a change in the growth intensity of the Staphylococcus aureus colony between these two points.
  The collected material was placed in a test-tube with a transport medium and transferred to the laboratory of the University Children's Hospital in Lublin, where it was inoculated on appropriate media. Microbial growth was assessed by semi-quantitative method (+ scanty growth, ++ moderate growth, +++ large growth, ++++ abundant growth).

SECONDARY OUTCOMES:
Incidence of treatment emergent adverse events [safety and tolerability] | from baseline, up to the 3-month time point
  Incidence, frequency and severity of treatment emergent adverse events.
Incidence of treatment emergent adverse events leading to discontinuation [safety and tolerability] | from baseline, up to the 3-month time point
  The number of participants with adverse events leading to discontinuation.
Time to discontinuation due to treatment emergent adverse events [safety and tolerability] | From date of randomization until the date of occurrence of an adverse event leading to discontinuation, assessed up to 3 months
  To assess the time that has elapsed since treatment initiation to the occurrence of an adverse event leading to discontinuation.
Incidence of treatment emergent abnormalities in physical examination findings [safety and tolerability] | at baseline, and at 3-months
  Observe skin, lymph nodes, ears, eyes, nose, throat, cardiac and pulmonary status, abdomen and extremities for any abnormalities.
Incidence of treatment emergent abnormalities in pulse rate [safety and tolerability] | at baseline, and at 3-months
  Measure resting pulse rate as beats per minute.
Incidence of treatment emergent abnormalities in blood pressure [safety and tolerability] | at baseline, and at 3-months
  Measure systolic and diastolic blood pressure (in mmHg).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pulmonary Diseases and Children Rheumatology, Medical University of Lublin, Lublin, Poland

REFERENCES:
- [Background] Janeczek K, Emeryk A, Rachel M, Duma D, Zimmer L, Poleszak E. Polyvalent Mechanical Bacterial Lysate Administration Improves the Clinical Course of Grass Pollen-Induced Allergic Rhinitis in Children: A Randomized Controlled Trial. J Allergy Clin Immunol Pract. 2021 Jan;9(1):453-462. doi: 10.1016/j.jaip.2020.08.025. Epub 2020 Aug 26. PMID 32858239
- [Background] Janeczek KP, Emeryk A, Rapiejko P. Effect of polyvalent bacterial lysate on the clinical course of pollen allergic rhinitis in children. Postepy Dermatol Alergol. 2019 Aug;36(4):504-505. doi: 10.5114/ada.2019.87457. Epub 2019 Aug 30. No abstract available. PMID 31616231
- [Background] Banche G, Allizond V, Mandras N, Garzaro M, Cavallo GP, Baldi C, Scutera S, Musso T, Roana J, Tullio V, Carlone NA, Cuffini AM. Improvement of clinical response in allergic rhinitis patients treated with an oral immunostimulating bacterial lysate: in vivo immunological effects. Int J Immunopathol Pharmacol. 2007 Jan-Mar;20(1):129-38. doi: 10.1177/039463200702000115. PMID 17346436
- [Background] Meng Q, Li P, Li Y, Chen J, Wang L, He L, Xie J, Gao X. Broncho-vaxom alleviates persistent allergic rhinitis in patients by improving Th1/Th2 cytokine balance of nasal mucosa. Rhinology. 2019 Dec 1;57(6):451-459. doi: 10.4193/Rhin19.161. PMID 31403136
- [Background] Han L, Zheng CP, Sun YQ, Xu G, Wen W, Fu QL. A bacterial extract of OM-85 Broncho-Vaxom prevents allergic rhinitis in mice. Am J Rhinol Allergy. 2014 Mar-Apr;28(2):110-6. doi: 10.2500/ajra.2013.27.4021. PMID 24717947
- [Background] Liu C, Huang R, Yao R, Yang A. The Immunotherapeutic Role of Bacterial Lysates in a Mouse Model of Asthma. Lung. 2017 Oct;195(5):563-569. doi: 10.1007/s00408-017-0003-8. Epub 2017 May 4. PMID 28474108
- [Background] Esposito S, Soto-Martinez ME, Feleszko W, Jones MH, Shen KL, Schaad UB. Nonspecific immunomodulators for recurrent respiratory tract infections, wheezing and asthma in children: a systematic review of mechanistic and clinical evidence. Curr Opin Allergy Clin Immunol. 2018 Jun;18(3):198-209. doi: 10.1097/ACI.0000000000000433. PMID 29561355
- [Background] Emeryk A, Bartkowiak-Emeryk M, Raus Z, Braido F, Ferlazzo G, Melioli G. Mechanical bacterial lysate administration prevents exacerbation in allergic asthmatic children-The EOLIA study. Pediatr Allergy Immunol. 2018 Jun;29(4):394-401. doi: 10.1111/pai.12894. PMID 29575037
- [Background] Refaat MM, Ahmed TM, Ashour ZA, Atia MY. Immunological role of nasal staphylococcus aureus carriage in patients with persistent allergic rhinitis. Pan Afr Med J. 2008 Oct 30;1:3. PMID 21532892
- [Background] Hohchi N, Hashida K, Ohkubo J, Wakasugi T, Mori T, Nguyen KH, Kuroda E, Ikeno T, Taniguchi H, Suzuki H. Synergism of Staphylococcus aureus colonization and allergic reaction in the nasal cavity in mice. Int Arch Allergy Immunol. 2012;159(1):33-40. doi: 10.1159/000335200. Epub 2012 May 3. PMID 22555155
- [Background] Cevik C, Yula E, Yengil E, Gulmez MI, Akbay E. Identification of nasal bacterial flora profile and carriage rates of methicillin-resistant Staphylococcus aureus in patients with allergic rhinitis. Eur Arch Otorhinolaryngol. 2014 Jan;271(1):103-7. doi: 10.1007/s00405-013-2492-2. Epub 2013 Apr 17. PMID 23591798
- [Background] Shiomori T, Yoshida S, Miyamoto H, Makishima K. Relationship of nasal carriage of Staphylococcus aureus to pathogenesis of perennial allergic rhinitis. J Allergy Clin Immunol. 2000 Mar;105(3):449-54. doi: 10.1067/mai.2000.104256. PMID 10719292
- [Background] Zagolski O, Strek P, Kasprowicz A, Bialecka A. Effectiveness of Polyvalent Bacterial Lysate and Autovaccines Against Upper Respiratory Tract Bacterial Colonization by Potential Pathogens: A Randomized Study. Med Sci Monit. 2015 Oct 5;21:2997-3002. doi: 10.12659/MSM.893779. PMID 26434686
- [Result] Janeczek K, Emeryk A, Zimmer L, Poleszak E, Ordak M. Nasal carriage of Staphylococcus aureus in children with grass pollen-induced allergic rhinitis and the effect of polyvalent mechanical bacterial lysate immunostimulation on carriage status: A randomized controlled trial. Immun Inflamm Dis. 2022 Mar;10(3):e584. doi: 10.1002/iid3.584. Epub 2021 Dec 29. PMID 34965026